CLINICAL TRIAL: NCT00249730
Title: A Prospective Multicenter, Parallel Group Study With A Single Blind Phase And A Double Blind Randomised Phase, To Evaluate The Efficacy And Satisfaction Of Viagra (Sildenafil Citrate) High Dose (100mg) Titration Compared With 50mg Dose, In Men With Erectile Dysfunction
Brief Title: Titration Study to Evaluate Efficacy and Satisfaction of Viagra in Men With Erectile Function.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A1481237
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Impotence
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

INTERVENTIONS:
Drug: Sildenafil

SUMMARY:
To evaluate the efficacy of Viagra dose titration to 100mg versus 50mg in men with erectile dysfunction, based on responses to the IIEF questionnaire as measured at the beginning and at the end of double blind treatment, comparing the group titrated to 100mg vs. the group maintained on 50mg.

ELIGIBILITY:
Inclusion Criteria:

* Documented clinical diagnosis of ED by using IIEF-EF domain with score of â‰¤ 25.
* Subjects must be in a stable relationship with the same partner for at least 6 months and willing to attempt sexual intercourse.

Exclusion Criteria:

* Subjects in whom sexual activity is inadvisable in the opinion of the investigator such as significant cardiovascular disease in the last 6 months; including cardiac failure, myocardial infarction, unstable angina, stroke or transient ischemic attack (TIA), symptomatic or clinically significant cardiac arrhythmias including atrial fibrillation.
* Subjects who are currently taking or are likely to be treated with nitrates or nitric oxide donors in any form (oral, sublingual, buccal, transdermal, inhalational or as aerosols) on either regular or intermittent basis.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510
Dates: Start 2005-10

PRIMARY OUTCOMES:
Change in IIEF erectile function domain score at the end of double blind treatment.

SECONDARY OUTCOMES:
Change in other IIEF domain scores; Response to other questionnaires regarding treatment satisfaction, safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- Canada (5):
  - Pfizer Investigational Site, Kitchener, Ontario
  - Pfizer Investigational Site, Sarnia, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Saint-Léonard, Quebec
  - Pfizer Investigational Site, Trois-Rivières, Quebec
- France (4):
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
- Greece (3):
  - Pfizer Investigational Site, Goudi, Athens
  - Pfizer Investigational Site, Pátrai
  - Pfizer Investigational Site, Thessaloniki
- Israel (4):
  - Pfizer Investigational Site, Beersheba
  - Pfizer Investigational Site, Haifa
  - Pfizer Investigational Site, Petah Tikva
  - Pfizer Investigational Site, Tel Aviv
- Italy (5):
  - Pfizer Investigational Site, Bologna
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, L’Aquila
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Roma
- Pfizer Investigational Site, Moscow, Russia
- Spain (7):
  - Pfizer Investigational Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Pfizer Investigational Site, Alicante
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Málaga
  - Pfizer Investigational Site, Seville
  - Pfizer Investigational Site, Valencia
- United Kingdom (10):
  - Pfizer Investigational Site, Belmont, Durham
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Weybridge, Surrey
  - Pfizer Investigational Site, Chippenham, Wilts.
  - Pfizer Investigational Site, Trowbridge, Wiltshire
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Doncaster
  - Pfizer Investigational Site, Dundee
  - Pfizer Investigational Site, Glasgow

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481237&StudyName=Titration+study+to+evaluate+efficacy+and+satisfaction+of+Viagra+in+men+with+erectile+function%2E